CLINICAL TRIAL: NCT00981916
Title: Ultrasound Determination of Needle Depth in Lumbar and Thoracic Epidurals in Adult Non-Parturient Patients
Brief Title: Ultrasound Determination of Needle Depth in Epidurals in Adult Patients
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 16451A
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Analgesia, Epidural; Surgery
Keywords: determination of depth to epidural space using ultrasound
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The introduction of local anesthetics and other medications into the epidural space is a principal technique in provision of anesthesia in many procedures. Typically the anesthetist accesses the epidural space blindly using palpation and visualization of external landmarks and then uses a needle to get to the epidural space. The investigators propose a prospective study of use of ultrasound in a large heterogeneous group of surgical candidates to define the relationship between the actual needle depth (ND) to the epidural space and measured ultrasound depth (UD). Establishing correctly the depth to the epidural space via ultrasound is a component of ultrasound imaging that might improve current technique, and might lead to faster performance of the epidural. Use of ultrasound may also improve the efficacy and safety of epidural placement.

The null hypothesis of this study is that ultrasound depth is similar to the needle depth in adult non parturient patients undergoing lumbar and thoracic epidurals. A parturient in this case is defined as a female currently near or going through labor.

ELIGIBILITY:
Inclusion Criteria:

* The patient population will include all non parturients above the age of 18 who are candidates for epidural placement prior to surgery.

Exclusion Criteria:

* Parturients, prisoners and patients younger than 18 years old will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population will include all non parturients above the age of 18 who are candidates for epidural placement prior to surgery
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Ultrasound depth | At time of exam
  Depth to epidural space as determined by ultrasound probe

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago, Chicago, Illinois, United States